CLINICAL TRIAL: NCT01643889
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Single- and Multiple-Dose, 4-Way Crossover Study to Evaluate the Effects of Domperidone on Cardiac Repolarization in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Domperidone on Cardiac Repolarization in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR100893; DOMDYP1001 (Other: Janssen Research & Development, LLC); 2012-001567-70 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; Domperidone; Cardiac Repolarization
MeSH Terms: interventions — Domperidone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Sequence group ADBC (Experimental): Treatment A: domperidone 10 mg; Treatment B: domperidone 20 mg; Treatment C: placebo; Treatment D: moxifloxacin.
  Interventions: Drug: Treatment A (domperidone 10 mg); Drug: Treatment B (domperidone 20 mg); Drug: Treatment C (placebo); Drug: Treatment D (moxifloxacin)
- Sequence group BACD (Experimental): Treatment A: domperidone 10 mg; Treatment B: domperidone 20 mg; Treatment C: placebo; Treatment D: moxifloxacin.
  Interventions: Drug: Treatment A (domperidone 10 mg); Drug: Treatment B (domperidone 20 mg); Drug: Treatment C (placebo); Drug: Treatment D (moxifloxacin)
- Sequence group CBDA (Experimental): Treatment A: domperidone 10 mg; Treatment B: domperidone 20 mg; Treatment C: placebo; Treatment D: moxifloxacin.
  Interventions: Drug: Treatment A (domperidone 10 mg); Drug: Treatment B (domperidone 20 mg); Drug: Treatment C (placebo); Drug: Treatment D (moxifloxacin)
- Sequence group DCAB (Experimental): Treatment A: domperidone 10 mg; Treatment B: domperidone 20 mg; Treatment C: placebo; Treatment D: moxifloxacin.
  Interventions: Drug: Treatment A (domperidone 10 mg); Drug: Treatment B (domperidone 20 mg); Drug: Treatment C (placebo); Drug: Treatment D (moxifloxacin)

INTERVENTIONS:
Drug: Treatment A (domperidone 10 mg) — 1 domperidone 10 mg capsule four times a day (q.i.d.) + 1 domperidone placebo capsule q.i.d. on Days 1 to 3 and a single dose on Day 4 (13 doses in total), and 1 moxifloxacin placebo capsule in the morning of Day 1.
Drug: Treatment B (domperidone 20 mg) — 2 domperidone 10 mg capsules four times a day (q.i.d.) on Days 1 to 3 and a single dose on Day 4 (13 doses in total), and 1 moxifloxacin placebo capsule in the morning of Day 1.
Drug: Treatment C (placebo) — 2 domperidone placebo capsules four times a day (q.i.d.) on Days 1 to 3 and a single dose on Day 4 (13 doses in total), and 1 moxifloxacin placebo capsule in the morning of Day 1.
Drug: Treatment D (moxifloxacin) — 2 domperidone placebo capsules four times a day (q.i.d.) on Days 1 to 3 and a single dose on Day 4 (13 doses in total), and 1 moxifloxacin 400 mg capsule in the morning of Day 1.

SUMMARY:
The purpose of this study is to assess the effects of single and multiple doses of domperidone on the QTc interval duration in healthy adult volunteers at domperidone doses of 10 mg four times a day (q.i.d.) and 20 mg q.i.d.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), placebo- and positive-controlled, double-blind (neither physician nor participant knows the treatment that the participant receives), single-dose and multiple-dose, 4-way crossover (method used to switch participants from one treatment arm to another in a clinical trial) study. A placebo control will be used to evaluate the effect of domperidone on QTc intervals in comparison with placebo. QTc is a measure of time in the heart electrical cycle. Placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial. Moxifloxacin, which is known to prolong QTc intervals, will be used as positive control to establish assay sensitivity. The participants will be randomly assigned to 1 of 4 treatment sequence groups (ADBC, BACD, CBDA, and DCAB) based on a computer-generated randomization schedule and will receive the following 4 treatments in the order specified by the randomization: Treatment A (10 mg domperidone); Treatment B (20 mg domperidone); Treatment C (placebo); Treatment D (moxifloxacin). The study has 3 phases: a screening phase, a double-blind treatment phase (that corresponds to 4 treatment periods), and an assessment period. Each treatment period will last 4 days and will be separated with a washout period (ie, period when receiving no treatment) of 4 to 9 days. The participants will be confined to the clinical testing facility for approximately 5 days in each period. All treatments (A, B, C and D) will be given orally with water. The maximum study duration for a participant will be 74 days.

ELIGIBILITY:
Inclusion Criteria:

* If a woman, must be postmenopausal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control
* If a woman, must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day -1 of each treatment period
* Body mass index (BMI; weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* An electrocardiogram (ECG) consistent with normal cardiac conduction and function

Exclusion Criteria:

* History of risk factors for cardiac diseases
* Laboratorial tests with clinically significant abnormal values
* Clinically significant abnormal physical examination, vital signs or electrocardiogram (ECG) at screening
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol within 14 days before the first dose of the study drug
* History of or current clinically significant medical illness, disease, or condition that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The change from baseline in QTc intervals on Day 1 | Baseline, 5 hours
The change from baseline in QTc intervals on Day 4 | Baseline, 5 hours

SECONDARY OUTCOMES:
The plasma concentrations of domperidone | 9 time points on Day 1
The plasma concentrations of domperidone | 9 time points on Day 4
The plasma concentrations of moxifloxacin | 9 time points on Day 1
The plasma concentrations of moxifloxacin | 9 time points on Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Single- and Multiple-Dose, 4-Way Crossover Study to Evaluate the Effects of Domperidone on Cardiac Repolarization in Healthy Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3561&filename=CR100893_CSR.pdf